CLINICAL TRIAL: NCT03287999
Title: Inter Individual Variability in Initiation Pathway Activation and Regulation and Phenotypic Heterogeneity in Patients With Haemophilia A and B
Acronym: InPath
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Pratima Chowdary, Dr Pratima Chowdary, Royal Free Hospital NHS Foundation Trust
Other Study IDs: 11296
Record Dates: First submitted 2017-09-13; First posted 2017-09-19 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Haemophilia patients: Persons with haemophilia A or B - 240 to be recruited
  Interventions: Diagnostic Test: Thrombophilia screen; Diagnostic Test: Initiation pathway analysis
- Healthy volunteers: Healthy volunteers - 10 to be recruited
  Interventions: Diagnostic Test: Thrombophilia screen; Diagnostic Test: Initiation pathway analysis

INTERVENTIONS:
Diagnostic Test: Thrombophilia screen — Thrombophilia screen (including antithrombin activity (AT:Ac), protein S antigen (PS:free), protein C activity (PC:Ac) , genetic analysis for FV Leiden and Prothrombin 3'UTR mutations and screening for lupus anticoagulant.
Diagnostic Test: Initiation pathway analysis — Evaluation of inter-individual variability in regulation of TF.VIIa.Xa.TFPI complex (tissue factor, activated Factor VII, activated factor X, tissue factor pathway inhibitor)

SUMMARY:
Severe haemophilia A and B (SHA, SHB) are X - linked inherited bleeding disorders, characterised by factor VIII and IX levels of <1 IU/dL respectively. The mainstay of treatment in SHA and SHB is replacement therapy with intravenous infusions of factor VIII and IX. However, there is significant variability in the bleeding phenotype within severe haemophiliacs with some presenting with minimal bleeding episodes even on less intensive treatment regimens. A significant contributor to inter-individual variability in the bleeding phenotype is the coagulation phenotype, but there are no established assays in routine clinical practice that can be used to quantify this. This study aims to study novel assays and characterise the observed phenotypic heterogeneity.

ELIGIBILITY:
Patients

Inclusion Criteria:

1. Patients with haemophilia A or B (baseline FVIII/FIX level <30%)
2. Age ≥ 18 years
3. Written informed consent in accordance with local and institutional guidelines.

Exclusion Criteria:

1. Patients currently enrolled into a clinical trial of investigational medicinal product for haemophilia.

Healthy Volunteers

Inclusion Criteria:

1. Currently not receiving any antiplatelet or anticoagulant therapy or other drugs that can affect the coagulation system.
2. Age ≥ 18 years
3. Written informed consent in accordance with local and institutional guidelines.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include patients severe or moderate haemophilia A or B who are currently attending study sites for routine follow up visits. In addition, 10 healthy volunteers will also be recruited to act as controls
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-10-02 (Estimated); Study Completion 2020-10-02 (Estimated)

PRIMARY OUTCOMES:
Initiation pathway correlation with clinical phenotype | Within 18 months of consent
  Correlate lab assays that characterise initiation pathway with clinical phenotype.

SECONDARY OUTCOMES:
Correlation analysis between FVIII:C/FIX:C levels and whole blood clotting time, thrombin generation in platelet poor plasma. | Within 18 months of consent
Evaluation the sensitivity and specificity of global assays for disease severity and clinical phenotype. | Within 18 months of consent
Correlation analysis between activation threshold of initiation pathway to thrombin generation and clinical phenotype | Within 18 months of consent

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Chowdary, Principal Investigator — Royal Free Hospitals NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No